CLINICAL TRIAL: NCT04973189
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Intravenous Administration of SHR-1707 in Healthy Young Adult and Elderly Subjects
Brief Title: A Study of SHR-1707 in Healthy Young Adult and Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SHR-1707-101
Record Dates: First submitted 2021-06-08; First posted 2021-07-22 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: SHR-1707 compared with placebo
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A single dose of SHR-1707 by intravenous infusion in healthy young adults. (Experimental)
  Interventions: Drug: SHR-1707
- placebo in healthy young adults. (Placebo Comparator)
  Interventions: Drug: Placebo
- A single dose of SHR-1707 by intravenous infusion in elderly subjects. (Experimental)
  Interventions: Drug: SHR-1707
- placebo in elderly subject (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-1707 — A single dose of SHR-1707 by intravenous (IV) infusion in healthy young adults.
  Arms: A single dose of SHR-1707 by intravenous infusion in healthy young adults.
Drug: Placebo — A single dose of matching SHR-1707 placebo by intravenous (IV) infusion in healthy young adults.
  Arms: placebo in healthy young adults.
Drug: SHR-1707 — A single dose of SHR-1707 by intravenous (IV) infusion in elderly subjects.
  Arms: A single dose of SHR-1707 by intravenous infusion in elderly subjects.
Drug: Placebo — A single dose of matching SHR-1707 placebo by intravenous (IV) infusion in elderly subjects.
  Arms: placebo in elderly subject

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single intravenous administration of SHR-1707 in healthy young adult and elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures and possible adverse events, be able and willing to provide a written informed consent
2. Male or female aged between 18 years and 45 years (inclusive) at the date of signed consent form in Part 1 and aged between 55 years and 80 years (inclusive) in Part 2
3. Total body weight of 45~100 kg (inclusive), with a body mass index (BMI) of 19~28 kg/m2 (inclusive)
4. Subjects with good general health, no clinically significant abnormalities, or have underlying disease which is believed to have minimal impact on the study treatment in elderly subjects
5. WOCBP agree to take effective contraceptive methods

Exclusion Criteria:

1. Severe injuries or surgeries within 6 months before screening
2. Positive hepatitis B virus (HBsAg), hepatitis C virus (HCV-Ab), or human immunodeficiency virus (HIV-Ab) at screening
3. ALT, or AST or total bilirubin level <1.5x upper limit of normal range (ULN) at screening or baseline visits
4. QTcF > 450msec (Male), QTcF > 470msec (Female) in 12-lead ECG test during screening and baseline
5. Known history or suspected of being allergic to Aβ antibody
6. Use of any medicine within 14 days (including any prescription, or over-the-counter medicine, herbal remedy or nutritional supplement, except for vitamins and acetaminophen with recommended dose [The dose of acetaminophen should be less than 2g/day, and no more than 3 days for continuous use]), or within 5 half-lives
7. Live (attenuated) vaccination within 1 month before screening
8. Blood donation or loss of more than 400 mL of blood within 3 months; or received blood transfusion within 3 months before screening.
9. History of alcohol abuse in the past 12 months of screening
10. History of illicit or prescription drug abuse or addiction within 12 months of screening
11. More than 5 cigarettes daily for 12 months before screening
12. Participation in clinical trials of other investigational drugs (include placebo) or medical devices within 3 months prior to screening
13. Researchers and relevant staff of the research center or other persons directly involved in the implementation of the program
14. The instigators determined that other conditions were inappropriate for participation in this clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-05-08 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events as a Measure of Safety and Tolerability | Start of Treatment to end of study (approximately 12 weeks)
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Area under the concentration-time curve from time 0 to last time point (AUC0-last) after SHR-1707 administration | Start of Treatment to end of study (approximately 12 weeks)
  Area under the concentration-time curve from time 0 to last time point after SHR-1707 administration
Area under the concentration-time curve from time 0 to infinity (AUC0-inf) after SHR-1707 administration | Start of Treatment to end of study (approximately 12 weeks)
  Area under the concentration-time curve from time 0 to infinity after SHR-1707 administration
Time to Cmax (Tmax) of SHR-1707 | Start of Treatment to end of study (approximately 12 weeks)
  Time to Cmax of SHR-1707
Maximum observed concentration (Cmax) of SHR-1707 | Start of Treatment to end of study (approximately 12 weeks)
  Maximum observed concentration of SHR-1707
Terminal elimination half-life (t1/2) of SHR-1707 | Start of Treatment to end of study (approximately 12 weeks)
  Terminal elimination half-life of SHR-1707
Clearance (CL) of SHR-1707 | Start of Treatment to end of study (approximately 12 weeks)
  Clearance of SHR-1707
Volume of distribution (Vss) of SHR-1707 | Start of Treatment to end of study (approximately 12 weeks)
  Volume of distribution of SHR-1707
Mean residence time (MRT) of SHR-1707 | Start of Treatment to end of study (approximately 12 weeks)
  Mean residence time of SHR-1707
The change from baseline in plasma Aβ40 and Aβ42 concentrations | Start of Treatment to end of study (approximately 12 weeks)
  The change from baseline in plasma Aβ40 and Aβ42 concentrations will be measured to determine the degree of change over time.
Number of subjects with Anti-SHR-1707 antibodies | Start of Treatment to end of study (approximately 12 weeks)
  Number of subjects with positive ADA titers over time for SHR-1707

CONTACTS AND LOCATIONS:
Locations (1):
- The second Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang Y, Qiu H, Fan Y, Zhang Q, Qin H, Wu J, Zhang X, Liu Y, Zhou R, Zhang Q, Ye Z, Ma J, Xu Y, Feng S, Fei Y, Li N, Cui X, Dong F, Wang Q, Shen K, Shakib S, Williams J, Hu W. Safety, tolerability, pharmacokinetics and pharmacodynamics of a single intravenous dose of SHR-1707 in healthy adult subjects: two randomized, double-blind, single-ascending-dose, phase 1 studies. Alzheimers Res Ther. 2024 Oct 10;16(1):218. doi: 10.1186/s13195-024-01584-8. PMID 39390616